CLINICAL TRIAL: NCT03722641
Title: A Randomized, Single-blind, Crossover Study to Evaluate Postprandial Glycaemia in a Healthy Population After Intake of Milk and Oat Based Products
Brief Title: Evaluation of Postprandial Glycaemia in a Healthy Population After Intake of Milk and Oat Based Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TR1801
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-10

CONDITIONS: Healthy
MeSH Terms: interventions — Ornithine-Oxo-Acid Transaminase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Bread reference (Placebo Comparator): A standardized (50 grams carbohydrates) breakfast meal will be provided based on bread.
  Interventions: Other: Bread reference; Other: Product 1: Milk; Other: Product 2: Full fat milk + oat; Other: Product 3: Skim milk + oat, high fibre; Other: Product 4: Skim milk + oat, low fibre
- Product 1: Milk (Experimental): A standardized (50 grams carbohydrates) breakfast meal will be provided based on bread and a test product based on milk.
  Interventions: Other: Bread reference; Other: Product 1: Milk; Other: Product 2: Full fat milk + oat; Other: Product 3: Skim milk + oat, high fibre; Other: Product 4: Skim milk + oat, low fibre
- Product 2: Full fat milk + oat (Experimental): A standardized (50 grams carbohydrates) breakfast meal will be provided based on bread and a test product based on full fat milk and oat with high fiber content.
  Interventions: Other: Bread reference; Other: Product 1: Milk; Other: Product 2: Full fat milk + oat; Other: Product 3: Skim milk + oat, high fibre; Other: Product 4: Skim milk + oat, low fibre
- Product 3: Skim milk + oat, high fibre (Experimental): A standardized (50 grams carbohydrates) breakfast meal will be provided based on bread and a test product based on skim milk and oat with high fiber content.
  Interventions: Other: Bread reference; Other: Product 1: Milk; Other: Product 2: Full fat milk + oat; Other: Product 3: Skim milk + oat, high fibre; Other: Product 4: Skim milk + oat, low fibre
- Product 4: Skim milk + oat, low fibre (Experimental): A standardized (50 grams carbohydrates) breakfast meal will be provided based on bread and a test product based on skim milk and oat with low fiber content.
  Interventions: Other: Bread reference; Other: Product 1: Milk; Other: Product 2: Full fat milk + oat; Other: Product 3: Skim milk + oat, high fibre; Other: Product 4: Skim milk + oat, low fibre

INTERVENTIONS:
Other: Bread reference — Commercially available white wheat bread
Other: Product 1: Milk — Developed reference product based on milk
Other: Product 2: Full fat milk + oat — Developed product based on full fat milk with addition of oat
Other: Product 3: Skim milk + oat, high fibre — Developed product based on skim milk with addition of oat giving a high fiber content to the product
Other: Product 4: Skim milk + oat, low fibre — Developed product based on skim milk with addition of oat giving a lower fiber content to the product

SUMMARY:
The objective of this study is to investigate the effect on postprandial glycaemia in a healthy population after intake of milk and oat based products.

DETAILED DESCRIPTION:
Postprandial glycaemia, insulinaemia and GLP-1 will be measured after intake of test meals with equal amount of carbohydrates (adjusted using bread) and equal amount of total water.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 20 to 40 years of age
2. BMI 20-27 (±0.5) kg/m²
3. Agree to maintain consistent dietary habits and physical activity levels for the duration of the study
4. Healthy as determined by medical history and information provided by the volunteer
5. Willingness to complete questionnaires and follow instructions associated with the study and to complete all visits
6. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Elevated fasting blood glucose (at or above 6.1 mmol/L at fasting on visit 2, 3, 4 or 5)
2. Elevated fasting insulin (above 25 mIE/L)
3. Women who are pregnant or breast feeding
4. Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the SI
5. Use of medication, over-the-counter medication, natural health products or dietary supplements/probiotics that may affect glucose metabolism is prohibited during this study. Significance to be assessed by the SI. Participants who are taking allowed prescribed medications must agree to maintain their current method and dosing regimen during the course of the study unless recommended by their physician.
6. Known Type I or Type II diabetes, including women who previously have had gestational diabetes.
7. Use of antibiotics within 2 weeks of enrollment
8. Metabolic diseases and/or chronic gastrointestinal diseases (IBS, Crohns etc.)
9. Allergy to ingredients included in investigational product, placebo or standardized meal
10. Participants restricted to a vegetarian or vegan diet
11. Intolerance to lactose or gluten
12. Individuals who are averse to venous catheterization or capillary blood sampling
13. Currently active smokers (or using other tobacco products, and e-cigarettes)
14. Unstable medical conditions as determined by SI
15. Participation in other clinical research trials
16. Individuals who are cognitively impaired and/or who are unable to give informed consent
17. Acute infection
18. Any other condition which in the SI's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemia capillary | 0-120 min after consumption
  Primary outcome is the difference in the two-hour incremental area under the curve (iAUC (0 - 120 min)) for capillary blood glucose between product 1-4 and the bread reference.

SECONDARY OUTCOMES:
Postprandial glycaemia intravenous | 0-120 min
  The difference in the two-hour iAUC (0 - 120 min) for intravenous blood glucose between product 1-4 and the bread reference.
Postprandial Cmax capillary glucose | 0-180 min
  The difference in the three-hour Cmax (0 - 180 min) of capillary blood glucose between product 1-4 and the bread reference.
Postprandial Cmax venous glucose | 0-180 min
  The difference in the three-hour Cmax (0 - 180 min) of intravenous blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia capillary | 0-180 min
  The difference in the three-hour iAUC (0 - 180 min) of capillary blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia venous | 0-180 min
  The difference in the three-hour iAUC (0 - 180 min) of intravenous blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia capillary | 0-60 min
  The difference in the one-hour iAUC (0 - 60 min) of capillary blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia venous | 0-60 min
  The difference in the one-hour iAUC (0 - 60 min) of intravenous blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia Tmax capillary | 0-180 min
  The difference in the Tmax (the time to maximum concentration) of capillary blood glucose between product 1-4 and the bread reference.
Postprandial glycaemia Tmax venous | 0-180 min
  The difference in the Tmax of intravenous blood glucose between product 1-4 and the bread reference.
Postprandial insulinaemia | 0-180 min
  The difference in the three-hour iAUC (0 - 180 min) of intravenous blood insulin between product 1-4 and the bread reference.
Postprandial insulinaemia | 0-120 min
  The difference in the two-hour iAUC (0 - 120 min) of intravenous blood insulin between product 1-4 and the bread reference.
Postprandial insulinaemia | 0-60 min
  The difference in the one-hour iAUC (0 - 60 min) of intravenous blood insulin between product 1-4 and the bread reference.
Postprandial insulinaemia Cmax | 0-180 min
  The difference in the three-hour Cmax (0 - 180 min) of intravenous blood insulin between product 1-4 and the bread reference.
Postprandial insulinaemia Tmax | 0-180 min
  The difference in the Tmax of intravenous blood insulin between product 1-4 and the bread reference.
Postprandial GLP-1 bread reference | 0-60 min
  The difference in the one-hour iAUC (0 - 60 min) of intravenous blood GLP-1 between product 1-4 and the bread reference.
Postprandial GLP-1, yoghurt control | 0-60 min
  The difference in the one-hour iAUC (0 - 60 min) of intravenous blood GLP-1 between products 2-4 and product 1.
Postprandial GLP-1 Cmax bread reference | 0-60 min
  The difference in the one-hour Cmax (0 - 60 min) of intravenous blood GLP-1 between product 1-4 and the bread reference.
Postprandial GLP-1 Cmax yoghurt control | 0-60 min
  The difference in the one-hour Cmax (0 - 60 min) of intravenous blood GLP-1 between products 2-4 and product 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Aventure AB, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No